CLINICAL TRIAL: NCT04479345
Title: Knowledge, Attitude and Practice of Gastrointestinal Endoscopists Toward PPE in COVID-19 Era
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidi Karam, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: COVID endoscopy
Record Dates: First submitted 2020-07-20; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Online questionnaire

SUMMARY:
Assessing the knowledge and practice of GIT endoscopists toward the use of PPE.

DETAILED DESCRIPTION:
An online questionnaire assessing the knowledge and practice of GIT endoscopists toward the use of PPE will be used.

ELIGIBILITY:
Inclusion Criteria:

* GIT endoscopists

Exclusion Criteria:

* Refuse to participate

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GIT endoscopists
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The knowledge and attitude toward PPE during endoscopy | 2 months
  Online questionnaire

IPD SHARING:
Plan to Share IPD: No